CLINICAL TRIAL: NCT02967419
Title: The Study of the Relationship Between TWEAK/Fn14, JAK/STAT3 and IDO in the Immune Microenvironment of Endometrium in Repeated Implantation Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ZhangTao (Other)
Responsible Party: Sponsor-Investigator, ZhangTao, postgraduate of Tongji Hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-023
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Repeated Implantation Failure
Keywords: Repeated Implantation Failure; TWEAK;Fn14;JAK/STAT3;Indoleamine 2,3-dioxygenase

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine, endometrium

GROUPS / COHORTS (2):
- RIF group: People who were diagnosed as repeated implantation failure after IVF-ET
  Interventions: Other: No Intervention
- Control group: People who had normal pregnancy
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study is to find out the possible relationship among TWEAK/Fn14, JAK/STAT3 and IDO as well as their roles in the dysfunction of immune micro-environment of endometrium in people diagnosed as repeated implantation failure after in vitro Fertilization-embryo transfer(IVF-ET).

We will use the technology of Western-blot and Immunohistochemistry to find out the relationship of the expression of TWEAK/Fn14, JAK/STAT3 and IDO in endometrium . Also, we will use technology of Western-blot and Immunohistochemistry to determine whether there are differences of the the expression of TWEAK/Fn14, JAK/STAT3 and IDO in endometrium between RIF group and control group.

DETAILED DESCRIPTION:
The purpose of this study is to find out the possible relationship among TWEAK/Fn14, JAK/STAT3 and IDO as well as their roles in the dysfunction of immune micro-environment of endometrium in people diagnosed as repeated implantation failure after in vitro Fertilization-embryo transfer(IVF-ET).

We will use the technology of Western-blot and Immunohistochemistry to find out the relationship of the expression of TWEAK/Fn14, JAK/STAT3 and IDO in endometrium . Also, we will use technology of Western-blot and Immunohistochemistry to determine whether there are differences of the the expression of TWEAK/Fn14, JAK/STAT3 and IDO in endometrium between RIF group and control group.

ELIGIBILITY:
Inclusion Criteria:

- Women who had a history of implantation failures in at least three consecutive IVF attempts, in which 1-2 embryos of high grade quality are transferred in each cycle without diagnosis of any specific cause of implantation failure.

Exclusion Criteria:

- antiphospholipid syndrome (APS), endocrine disorder (diabetes, thyroid dysfunction), genetic disorders, uterine malformations, or any current infections

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of RIF is determined when transferred embryos fail to implant following in at least three consecutive IVF attempts, in which 1-2 embryos of high grade quality are transferred in each cycle.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
TWEAK/Fn14, JAK/STAT3 and IDO in Endometrium measured by Western-blot | 11/20/2016-12/30/2017

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Tongji Medicine College, Tongji Hospital, Reproductive Medicine Center, Wuhan, China

REFERENCES:
- [Background] Ledee N, Petitbarat M, Chevrier L, Vitoux D, Vezmar K, Rahmati M, Dubanchet S, Gahery H, Bensussan A, Chaouat G. The Uterine Immune Profile May Help Women With Repeated Unexplained Embryo Implantation Failure After In Vitro Fertilization. Am J Reprod Immunol. 2016 Mar;75(3):388-401. doi: 10.1111/aji.12483. Epub 2016 Jan 18. PMID 26777262
- [Background] Ashkar AA, Black GP, Wei Q, He H, Liang L, Head JR, Croy BA. Assessment of requirements for IL-15 and IFN regulatory factors in uterine NK cell differentiation and function during pregnancy. J Immunol. 2003 Sep 15;171(6):2937-44. doi: 10.4049/jimmunol.171.6.2937. PMID 12960317
- [Background] Mariee N, Li TC, Laird SM. Expression of leukaemia inhibitory factor and interleukin 15 in endometrium of women with recurrent implantation failure after IVF; correlation with the number of endometrial natural killer cells. Hum Reprod. 2012 Jul;27(7):1946-54. doi: 10.1093/humrep/des134. Epub 2012 Apr 26. PMID 22537815
- [Background] Petitbarat M, Rahmati M, Serazin V, Dubanchet S, Morvan C, Wainer R, de Mazancourt P, Chaouat G, Foidart JM, Munaut C, Ledee N. TWEAK appears as a modulator of endometrial IL-18 related cytotoxic activity of uterine natural killers. PLoS One. 2011 Jan 7;6(1):e14497. doi: 10.1371/journal.pone.0014497. PMID 21249128
- [Background] Ledee N, Petitbarat M, Rahmati M, Dubanchet S, Chaouat G, Sandra O, Perrier-d'Hauterive S, Munaut C, Foidart JM. New pre-conception immune biomarkers for clinical practice: interleukin-18, interleukin-15 and TWEAK on the endometrial side, G-CSF on the follicular side. J Reprod Immunol. 2011 Mar;88(2):118-23. doi: 10.1016/j.jri.2011.01.007. Epub 2011 Feb 18. PMID 21334074
- [Background] Lei M, Qin L, Wang A, Jin Y, Zhao X, Qi X. Fn14 receptor appears as a modulator of ovarian steroid-related regulation of goat endometrial epithelial cell IL-18 expression. Am J Reprod Immunol. 2015 May;73(5):428-36. doi: 10.1111/aji.12343. Epub 2014 Nov 24. PMID 25421447
- [Background] Mas AE, Petitbarat M, Dubanchet S, Fay S, Ledee N, Chaouat G. Immune regulation at the interface during early steps of murine implantation: involvement of two new cytokines of the IL-12 family (IL-23 and IL-27) and of TWEAK. Am J Reprod Immunol. 2008 Apr;59(4):323-38. doi: 10.1111/j.1600-0897.2007.00567.x. PMID 18336386
- [Background] Petitbarat M, Serazin V, Dubanchet S, Wayner R, de Mazancourt P, Chaouat G, Ledee N. Tumor necrosis factor-like weak inducer of apoptosis (TWEAK)/fibroblast growth factor inducible-14 might regulate the effects of interleukin 18 and 15 in the human endometrium. Fertil Steril. 2010 Aug;94(3):1141-3. doi: 10.1016/j.fertnstert.2009.10.049. Epub 2009 Dec 11. PMID 20004376
- [Background] Chen W, Jin W, Hardegen N, Lei KJ, Li L, Marinos N, McGrady G, Wahl SM. Conversion of peripheral CD4+CD25- naive T cells to CD4+CD25+ regulatory T cells by TGF-beta induction of transcription factor Foxp3. J Exp Med. 2003 Dec 15;198(12):1875-86. doi: 10.1084/jem.20030152. PMID 14676299
- [Background] Hill M, Tanguy-Royer S, Royer P, Chauveau C, Asghar K, Tesson L, Lavainne F, Remy S, Brion R, Hubert FX, Heslan M, Rimbert M, Berthelot L, Moffett JR, Josien R, Gregoire M, Anegon I. IDO expands human CD4+CD25high regulatory T cells by promoting maturation of LPS-treated dendritic cells. Eur J Immunol. 2007 Nov;37(11):3054-62. doi: 10.1002/eji.200636704. PMID 17948274
- [Background] Brenk M, Scheler M, Koch S, Neumann J, Takikawa O, Hacker G, Bieber T, von Bubnoff D. Tryptophan deprivation induces inhibitory receptors ILT3 and ILT4 on dendritic cells favoring the induction of human CD4+CD25+ Foxp3+ T regulatory cells. J Immunol. 2009 Jul 1;183(1):145-54. doi: 10.4049/jimmunol.0803277. Epub 2009 Jun 17. PMID 19535644
- [Background] Ban Y, Chang Y, Dong B, Kong B, Qu X. Indoleamine 2,3-dioxygenase levels at the normal and recurrent spontaneous abortion fetal-maternal interface. J Int Med Res. 2013 Aug;41(4):1135-49. doi: 10.1177/0300060513487642. Epub 2013 Jul 11. PMID 23847296
- [Background] Zong S, Li C, Luo C, Zhao X, Liu C, Wang K, Jia W, Bai M, Yin M, Bao S, Guo J, Kang J, Duan T, Zhou Q. Dysregulated expression of IDO may cause unexplained recurrent spontaneous abortion through suppression of trophoblast cell proliferation and migration. Sci Rep. 2016 Jan 27;6:19916. doi: 10.1038/srep19916. PMID 26814137
- [Background] Obayashi Y, Ozaki Y, Goto S, Obayashi S, Suzumori N, Ohyama F, Tone S, Sugiura-Ogasawara M. Role of Indoleamine 2,3-Dioxygenase and Tryptophan 2,3-Dioxygenase in Patients with Recurrent Miscarriage. Am J Reprod Immunol. 2016 Jan;75(1):69-77. doi: 10.1111/aji.12434. Epub 2015 Oct 29. PMID 26511909
- [Background] Orabona C, Belladonna ML, Vacca C, Bianchi R, Fallarino F, Volpi C, Gizzi S, Fioretti MC, Grohmann U, Puccetti P. Cutting edge: silencing suppressor of cytokine signaling 3 expression in dendritic cells turns CD28-Ig from immune adjuvant to suppressant. J Immunol. 2005 Jun 1;174(11):6582-6. doi: 10.4049/jimmunol.174.11.6582. PMID 15905495
- [Background] Sun Y, Chin YE, Weisiger E, Malter C, Tawara I, Toubai T, Gatza E, Mascagni P, Dinarello CA, Reddy P. Cutting edge: Negative regulation of dendritic cells through acetylation of the nonhistone protein STAT-3. J Immunol. 2009 May 15;182(10):5899-903. doi: 10.4049/jimmunol.0804388. PMID 19414739
- [Background] Yu J, Wang Y, Yan F, Zhang P, Li H, Zhao H, Yan C, Yan F, Ren X. Noncanonical NF-kappaB activation mediates STAT3-stimulated IDO upregulation in myeloid-derived suppressor cells in breast cancer. J Immunol. 2014 Sep 1;193(5):2574-86. doi: 10.4049/jimmunol.1400833. Epub 2014 Jul 25. PMID 25063873
- [Background] Campia I, Buondonno I, Castella B, Rolando B, Kopecka J, Gazzano E, Ghigo D, Riganti C. An Autocrine Cytokine/JAK/STAT-Signaling Induces Kynurenine Synthesis in Multidrug Resistant Human Cancer Cells. PLoS One. 2015 May 8;10(5):e0126159. doi: 10.1371/journal.pone.0126159. eCollection 2015. PMID 25955018